CLINICAL TRIAL: NCT01797237
Title: Outcome Comparison Between PFNA and InterTAN in Intertrochanteric Fractures
Brief Title: Outcome Comparison Between PFNA and InterTAN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peifu Tang (Other)
Responsible Party: Sponsor-Investigator, Peifu Tang, Chief, Professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLAGH OD 14
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Intertrochanteric Fracture
Keywords: surgery; fixation; intramedullary nail
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stable intertrochanteric fracture (Experimental): The type of intertrochanteric fracture was below A2.1 (with A2.1) according to the AO/ATO classification.
  Interventions: Device: PFNA; Device: InterTAN
- Unstable intertrochanteric fracture (Experimental): The type of intertrochanteric fracture was above A2.1 (without A2.1) according to the AO/ATO classification.
  Interventions: Device: PFNA; Device: InterTAN

INTERVENTIONS:
Device: PFNA
  Other Names: Proximal Femoral Nail Antirotation (Synthes)
Device: InterTAN
  Other Names: InterTAN Femoral Nail (Smith&Nephew)

SUMMARY:
The purpose of this study is to determine whether this two intramedullary fixations are effectively in the treatment of intertrochanteric fracture.

DETAILED DESCRIPTION:
With the progress of aging society, elderly patients with intertrochanteric fractures were occurred more and more. The best recommend treatment is surgical treatment of intramedullary fixation. However, existing methods of intramedullary fixation could not be restored the integrated interior support, and it will occur early hip varus. Meanwhile, the varus deformity will no longer develop if the two ends contact with wach other. This new intramedullary fixation device can overcome the existing shortage of intramedullary fixation devices and supporting the inside of the problem. It can prompting the fracture site to obtain a stronger initial stability, improve fracture healing rate, reduce the incidence of varus and allow patients with early weight-bearing walking.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women aged 18 years and older (with no upper age limit).
* Fracture of the intertrochanteric fracture confirmed with either anteroposterior and lateral hip radiographs, computed tomography, or magnetic resonance imaging (MRI).
* Operative treatment of fractures within 14 days of presenting to the emergency room.
* Patient was ambulatory prior to fracture, though they may have used an aid such as a cane or a walker.
* Anticipated medical optimalization for operative fixation of the hip.
* Provision of informed consent by patient or legal guardian.
* No other major trauma.

Exclusion Criteria:

* Patients not suitable for internal fixation (i.e., severe osteoarthritis, rheumatoid arthritis, or pathologic fracture).
* Associated major injuries of the lower extremity (i.e., ipsilateral or contralateral fractures of the foot, ankle, tibia, fibula, knee, or femur; dislocations of the ankle, knee, or hip; or femoral head defects or fracture).
* Retained hardware around the affected hip.
* Infection around the hip (i.e., soft tissue or bone).
* Patients with disorders of bone metabolism except osteoporosis (i.e., Paget's disease, renal osteodystrophy, osteomalacia).
* Moderate or severe cognitively impaired patients (i.e., Six Item Screener with 3 or more errors).
* Patients with Parkinson's disease (or dementia) severe enough to increase the likelihood of falling or severe enough to compromise rehabilitation. Likely problems, in the judgment of the investigators, with maintaining follow-up. We will, for example, exclude patients with no fixed address, those who report a plan to move out of town in the next year, or intellectually challenged patients without adequate family support.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Quality of life | six months
  Assessment the quality of life by SF-36 (The Short Form Health Survey), ADL (Activities of Daily Living), FIM (Functional Independence Measure).

SECONDARY OUTCOMES:
Bone healing condition | Six months
  Bone healing condition was checked by radiological examination.

OTHER OUTCOMES:
Complications | Six months
  Death, implant breakage/failure, secondary fracture, infection and VTE (Venous Thromboembolism).

CONTACTS AND LOCATIONS:
Overall Officials: Peifu Tang, MD, Study Chair — Chinese PLA General Hospital; Lihai Zhang, MD, Study Director — Chinese PLA General Hospital; Qi Yao, MD, Principal Investigator — Beijing Shijitan Hospital, Capital Medical University; Wen Zhao, MD, Principal Investigator — Beijing Aerospace General Hospital
Locations (1):
- The General Hospital of the People's Liberation Army, Beijing, Beijing Municipality, China